CLINICAL TRIAL: NCT03693170
Title: Phase II, Open-label, Single Arm, Multicenter Study of Encorafenib, Binimetinib Plus Cetuximab in Subjects With Previously Untreated BRAF V600E -Mutant Metastatic Colorectal Cancer
Brief Title: Encorafenib, Binimetinib and Cetuximab in Subjects With Previously Untreated BRAF-mutant ColoRectal Cancer
Acronym: ANCHOR-CRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Pfizer (Industry); Merck KGaA, Darmstadt, Germany (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W00090 GE 2 01
Record Dates: First submitted 2018-09-17; First posted 2018-10-02 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: BRAF V600E-mutant Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; binimetinib; Cetuximab

STUDY DESIGN:
Masking Description: All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 Arm (Experimental): encorafenib plus binimetinib plus cetuximab
  Interventions: Drug: encorafenib; Drug: Binimetinib; Drug: Cetuximab

INTERVENTIONS:
Drug: encorafenib — 300 mg administered orally once daily (QD)
  Other Names: Braftovi
Drug: Binimetinib — Binimetinib 45 mg administered orally twice daily (BID)
  Other Names: Mektovi
Drug: Cetuximab — Standard of care for the 28 first weeks(*) and then every 2 weeks (**) :
  (*) 400 mg/m2 administered as a 120-min infusion on Cycle 1 Day 1, followed by 250 mg/m2 administered as a 60-min infusion once weekly (QW) for the first 28 weeks. (**) 500 mg/m2 administered as a 120-min infusion twice weekly (Q2W) from Week 29 (Cycle 8 Day 1) onward.
  Following implementation of an Urgent Safety Measure on 26 Mar 2020 due to the outbreak of COVID-19 pandemic, cetuximab infusions could be administered Q2W regardless of the cycle number, after investigator's evaluation of the benefit/risk ratio for the subject, with regards to COVID-19 pandemic.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the combination of study drugs encorafenib, binimetinib and cetuximab in patients who have BRAF V600 mutant metastatic colorectal cancer and have not received any prior treatment for their metastatic disease.

DETAILED DESCRIPTION:
The presence of a BRAFV600E mutation is considered a marker of poor prognosis in subjects with mCRC. The preclinical results and preliminary clinical data together justify the evaluation of this triple combination in the first-line setting of this population. The primary objective of the study is to evaluate the antitumor activity of the combination of encorafenib, binimetinib and cetuximab by assessing the overall response rate in adult subjects with previously untreated BRAFV600E-mutant metastatic colorectal cancer. It will also assess the effect of the triple combination on the duration of response, time to response, progression-free survival and overall survival and assess the effect on quality of life. It will also characterize the safety and tolerability of the triple combination as well as describe the pharmacokinetics (PK) of encorafenib, binimetinib, and cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Histologically or cytologically confirmed CRC that is metastatic
* Presence of BRAF V600E in tumor tissue determined by local assay at any time prior to screening
* Evidence of measurable disease as per RECIST, v1.1
* Subject able to receive cetuximab as per approved label with regards to RAS status
* Eastern Cooperative Oncology Group Status (ECOG) 0 or 1
* Adequate renal, hepatic, cardiac and bone marrow functions and adequate electrolytes as per protocol
* Subject able to take oral medications

Exclusion Criteria:

* Prior systemic therapy for metastatic disease
* Prior treatment with any RAF inhibitor, MEK inhibitor, cetuximab or other anti-EGFR inhibitors
* Symptomatic brain metastasis or Leptomeningeal disease
* History or current evidence of Retinal Vein Occlusion (RVO) or current risk factors for RVO
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤ 12 months prior to first dose.
* Impaired cardiovascular function or clinically significant cardiovascular diseases: history of myocardial infarction or coronary disorders within 6 months prior to start of study treatment, symptomatic congestive heart failure (grade 2 or higher), past or current clinically significant arrhythmia and/or conduction disorder within 6 months prior to study treatment start
* History of thromboembolic or cerebrovascular events within 6 months prior to start of study treatment
* Concurrent neuromuscular disorder that is associated with potential elevation of Creatine Kinase
* Known contraindication to cetuximab administration as per SPC/approved label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle KLAUCK, MD, Study Director — Corporate Medical&Patient/Consumer Division, Pierre Fabre Medicament
Locations (45):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - PC dba West Cancer Center, Germantown, Tennessee
- Krankenhaus der Barmherzigen Brüder, Vienna, Austria
- Belgium (3):
  - UZ Gent, Gastro-Enterology, Ghent, East Flanders
  - Trial DIO, UZ Gasthuisberg, Leuven, Flemish Brabant
  - Cliniques universitaires Saint-Luc, Brussels
- France (9):
  - ICM- VAL d 'Aurelle, Montpellier, Cedex 5
  - Hôpital Morvan CHRU de Brest Institut de cancérologie et d'hematologie, Brest
  - AP-HM CHU Timone, Marseille
  - Hôpital Cochin Gastroenterology, Paris
  - Hôpital Europeen Georges Pompidou, Paris
  - Hôpital Saint Antoine, Paris
  - HOPITAL HAUT-LEVEQUE, Av de MAGELLAN, Pessac
  - ICO- Site René Gauducheau, Saint-Herblain
  - CHU TOULOUSE Rangueil, Toulouse
- Italy (5):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Forlì-Cesena
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo
  - Ospedale Policlinic San Martin, Genova
  - Ospedale S.M. Misericordia, Perugia
- Japan (6):
  - Pierre Fabre Investigative Site, Nagoya, Aichi-ken
  - Pierre Fabre Investigative Site, Kashiwa, Chiba
  - Pierre Fabre Investigative Site, Fukuoka, Fukuoka
  - Pierre Fabre Investigative Site, Osaka, Osaka
  - Pierre Fabre Investigative Site, Nagaizumi-cho, Shizuoka
  - Pierre Fabre Investigative Site, Koto-ku,, Tokyo
- St Antonius Ziekenhuis, Utrecht, Netherlands
- Spain (12):
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Complejo Hospitalario De Navarra S Oncologia Medica, Pamplona, Navarre
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic I Provincial de Barcelona, Barcelona
  - Institut Català d'Oncologia (ICO L'Hospitalet), Barcelona
  - Hospital de la Santa Creu i Santa Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clínico Universitario de, Valencia
  - Hospital Universitario y Politécnico La FE, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Torbay Hospital, Lowes Bridge, Torquay, Devon
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James Hospital, Leeds
  - GI research team, OHCT, Guy's Hospital, London
  - GI Research Team, The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Van Cutsem E, Taieb J, Yaeger R, Yoshino T, Grothey A, Maiello E, Elez E, Dekervel J, Ross P, Ruiz-Casado A, Graham J, Kato T, Ruffinelli JC, Andre T, Carriere Roussel E, Klauck I, Groc M, Vedovato JC, Tabernero J. ANCHOR CRC: Results From a Single-Arm, Phase II Study of Encorafenib Plus Binimetinib and Cetuximab in Previously Untreated BRAFV600E-Mutant Metastatic Colorectal Cancer. J Clin Oncol. 2023 May 10;41(14):2628-2637. doi: 10.1200/JCO.22.01693. Epub 2023 Feb 10. PMID 36763936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 95 subjects were enrolled in the study between 17 January 2019 and 27 December 2019 in 68 investigational centers : 45 in EU, 7 in UK, 10 in USA and 6 in Japan
Pre-assignment Details: 125 subjects were screened for inclusion in the study. 30 subjects were excluded (29 due to eligibility criteria not met and 1 due to adverse event).
Groups:
- Encorafenib Plus Binimetinib Plus Cetuximab: Encorafenib: 300 mg QD. Binimetinib: 45 mg PO BID. Cetuximab: 400 mg/m2 intravenous (IV) at Cycle 1 day 1 then 250 mg/m2 (IV) every week (QW) for the first 28 weeks. Then, 500mg/m2 IV every two weeks (Q2W) from week 29 (Cycle 8 day 1)
Period: Overall Study
Arm/Group | Encorafenib Plus Binimetinib Plus Cetuximab
Started | 95
Completed | 20 (Participants with study treatment ongoing at the time of cut off date (29JUN2020))
Not Completed | 75
Not completed — Disease Progression | 48
Not completed — Adverse Event | 16
Not completed — Physician Decision | 6
Not completed — Protocol Violation | 2
Not completed — Death | 1
Not completed — Non compliance with study drug | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- 1 Arm: encorafenib plus binimetinib plus cetuximab
  encorafenib: Once daily, orally
  Binimetinib: Twice daily, orally
  Cetuximab: Standard of care for the 28 first weeks and then every 2 weeks
Arm/Group | 1 Arm
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [57 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 71
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 1
  Netherlands | 1
  Belgium | 9
  United States | 3
  Japan | 11
  Italy | 15
  United Kingdom | 13
  France | 13
  Spain | 29
Primary tumor location [Count of Participants; unit: Participants] — The category right-sided/transverse includes "Colon, Right " and "Colon, Transverse" tumor locations".
  The category left-sided includes "Colon, Left " and "Rectum" tumor locations".
  Participants
    Right-sided/transverse | 57
    Left-sided/rectum | 37
    Other | 1
Number of metastatic organs [Count of Participants; unit: Participants]
  1 | 23
  2 | 33
  >2 | 39
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. Scale is ranged from 0 to 5 with lower score meaning a lower functional impairment (0 corresponding to "fully active", 5 corresponding to death).
  Participants
    0 | 43
    1 | 52
Local BRAFV600E mutation result [Count of Participants; unit: Participants]
  Positive | 95
  Negative | 0
Central BRAFV600E mutation result [Count of Participants; unit: Participants]
  Positive | 92
  Negative | 2
  Indeterminate | 1
Metastatic organs [Count of Participants; unit: Participants]
  Adrenal gland | 3
  Bone | 4
  Liver | 52
  Lung | 35
  Lymph node | 49
  Mediastinum | 4
  Ovary | 3
  Peritoneum/Omentum | 46
  Pleural cavity | 3
  Rectum | 1
  Skin | 1
  Stomach | 2
  Other | 11
Prior antineoplastic therapy setting [Count of Participants; unit: Participants]
  Adjuvant | 17
  Neo-adjuvant | 3
  Locally advanced | 2
Prior antineoplastic monotherapy / combination [Count of Participants; unit: Participants]
  5-Fluorouracil + Folinic Acid | 4
  5-Fluorouracil + Folinic Acid + Oxaliplatin | 9
  Oxaliplatin + Capecitabine | 5
  Capecitabine | 6

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate (cORR) Based on Local Tumor Assessments
Description: The confirmed overall response rate (cORR) is the percentage of confirmed responses, defined as complete response (CR) or partial response (PR), as assessed by local radiologist/investigator review based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions; Partiel response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) = CR + PR.
Time Frame: From initiation of treatment to disease progression up to a maximum of 17.6 months.
Population: The Efficacy Set (ES) is composed of all included subjects having received at least one dose of study treatment (partial or full) with a centrally confirmed BRAFV600E mutation.
Measure: Number (95% Confidence Interval); unit: percentage of confirmed responses
Arm/Group | 1 Arm
Number analyzed (Participants) | 92
percentage of confirmed responses | 47.8 [37.3 to 58.5]
Statistical Analysis 1: Comparison: 1 Arm; The null hypothesis that the true response rate is 30% will be tested against a one-sided alternative. The cORR will be provided with a corresponding Clopper-Pearson (exact) binomial 95% CI for the Efficacy Set. This design yields a 1-sided type I error rate equal to 1.6% and power of 80% when the true response rate is 45%; Test type: Other; If 37 or more confirmed responses were observed in the 90 treated subjects with a centrally confirmed BRAFV600E mutation, corresponding to a lower limit of Clopper-Pearson (exact) binomial 95% CI exceeding 30%, the study was considered to have met its primary endpoint. If more than 90 subjects were enrolled, the lower limit of Clopper-Pearson was to be used for decision

2. Secondary Outcome: Confirmed Overall Response Rate (cORR) Based on Central Tumor Assessment
Description: The confirmed overall response rate (cORR) is the percentage of confirmed responses, defined as complete response (CR) or partial response (PR), as assessed by central radiologist review based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions; Partiel response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) = CR + PR.
Time Frame: From initiation of treatment to disease progression up to a maximum of 17.6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of confirmed responses
Groups:
- 1 Arm: encorafenib plus binimetinib plus cetuximab
  encorafenib: 300 mg administered orally once daily (QD)
  Binimetinib: Binimetinib 45 mg administered orally twice daily (BID)
  Cetuximab: Standard of care for the 28 first weeks(*) and then every 2 weeks (**) :
  (*) 400 mg/m2 administered as a 120-min infusion on Cycle 1 Day 1, followed by 250 mg/m2 administered as a 60-min infusion once weekly (QW) for the first 28 weeks. (**) 500 mg/m2 administered as a 120-min infusion twice weekly (Q2W) from Week 29 (Cycle 8 Day 1) onward.
  Following implementation of an Urgent Safety Measure on 26 Mar 2020 due to the outbreak of COVID-19 pandemic, cetuximab infusions could be administered Q2W regardless of the cycle number, after investigator's evaluation of the benefit/risk ratio for the subject, with regards to COVID-19 pandemic.
Arm/Group | 1 Arm
Number analyzed (Participants) | 92
percentage of confirmed responses | 45.7 [35.2 to 56.4]

3. Secondary Outcome: Overall Response Rate (ORR) Based on Local Tumor Assessments
Description: The overall response rate (ORR) is the percentage of responses, defined as complete response (CR) or partial response (PR), as assessed by local radiologist/investigator review based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions; Partiel response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) = CR + PR.
Time Frame: From initiation of treatment to disease progression up to a maximum of 17.6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responses
Arm/Group | 1 Arm
Number analyzed (Participants) | 92
percentage of responses | 62 [51.2 to 71.9]

4. Secondary Outcome: Overall Response Rate (ORR) Based on Central Tumor Assessments
Description: The overall response rate (ORR) is the percentage of responses, defined as complete response (CR) or partial response (PR), as assessed by central radiologist review based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions; Partiel response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) = CR + PR.
Time Frame: From initiation of treatment to disease progression up to a maximum of 17.6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responses
Arm/Group | 1 Arm
Number analyzed (Participants) | 92
percentage of responses | 60.9 [50.1 to 70.9]

5. Secondary Outcome: Duration of Response (DOR) Per Local Assessment
Description: Time from first radiographic evidence of response based on local radiologist/investigator review to the earliest documented PD or death due to underlying disease
Time Frame: From first radiographic evidence of response to disease progression up to a maximum of 17.6 months
Population: Confirmed responders per local radiologist/investigator assessment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 45
months | 5.1 [3.7 to 6.9]

6. Secondary Outcome: Duration of Response (DOR) Per Central Assessment
Description: Time from first radiographic evidence of response based on central review to the earliest documented PD or death due to underlying disease
Time Frame: From first radiographic evidence of response to disease progression up to a maximum of 17.6 months
Population: Confirmed responders per central assessment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 42
months | 5.1 [3.4 to 5.5]

7. Secondary Outcome: Time to Response (TTR) Per Local Review
Description: The TTR is defined as the time from the first dose until the first documented radiographic evidence of response of CR or PR per local review
Time Frame: From initiation of treatment to the first radiographic evidence of response up to a maximum of 17.6 months
Population: Confirmed responders per local radiologist/investigator assessment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 45
months | 1.4 [1.4 to 1.5]

8. Secondary Outcome: Time to Response (TTR) Per Central Review
Description: The TTR is defined as the time from the first dose until the first documented radiographic evidence of response of CR or PR per central review
Time Frame: From initiation of treatment to the first radiographic evidence of response up to a maximum of 17.6 months
Population: Confirmed responders per central assessment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 42
months | 1.4 [1.3 to 1.4]

9. Secondary Outcome: Progression-Free Survival (PFS) Per Local Review
Description: Time from first dose to the earliest documented date of disease progression based on local radiologist/investigator review or death due to any cause
Time Frame: From initiation of treatment to disease progression or death up to a maximum of 17.6 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 92
months | 5.8 [4.6 to 6.4]

10. Secondary Outcome: Progression of Free Survival (PFS) Per Central Review
Description: Time from first dose to the earliest documented date of disease progression based on central review or death due to any cause
Time Frame: From initiation of treatment to disease progression or death up to a maximum of 17.6 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 92
months | 5.0 [4.6 to 6.4]

11. Secondary Outcome: Overall Survival (OS)
Description: Time from first dose to death due to any cause
Time Frame: From initiation of treatment to death up to a maximum of 17.6 months
Population: The Full Analysis Set (FAS) is composed of all subjects having received at least one dose of study treatment (partial or full)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 Arm
Number analyzed (Participants) | 95
months | 17.2 [14.1 to NA] — Insufficient data maturity

12. Secondary Outcome: Plasma Concentration of Encorafenib
Description: Plasma concentration of encorafenib
Time Frame: 2 hours and 6 hours after dose on Day 1 cycle 1; Predose and 2 hours post dose on Day 1 cycle 2 (cycle length = 28 days)
Reporting Status: Not Posted

13. Secondary Outcome: Plasma Concentration of Binimetinib
Description: Plasma concentration of binimetinib
Time Frame: as for outcome 12
Reporting Status: Not Posted

14. Secondary Outcome: Plasma Concentration of Cetuximab
Description: Plasma concentration of cetuximab
Time Frame: as for outcome 12
Reporting Status: Not Posted

15. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Over Time
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for cancer subjects (EORTC QLQ-C30) includes a global health status/QoL. The scale ranges in score from 0 to 100, higher score on the global health status/QoL scale indicate higher QoL.
  Changes from baseline in EORTC QLQ-C30 global health status/quality of life (QoL) over time are presented in this record.
Time Frame: From Cycle 1 Day 1 (C1D1) Visit to the 30-day Safety Follow-up Visit up to a maximum of 17.6 months
Population: Changes from baseline are shown up to Cycle 10 Day 1 (C10D1) and for the 30-day safety follow-up period. Beyond C10D1, less than 10 subjects filled the questionnaire. Participants analyzed corresponds to the number of participant who completed the questionnaire the at the respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Arm
Number analyzed (Participants) | 95
units on a scale
  C2D1: number analyzed (Participants) | 79
  C2D1 | -2.64 (19.270)
  C3D1: number analyzed (Participants) | 71
  C3D1 | -0.35 (20.866)
  C4D1: number analyzed (Participants) | 69
  C4D1 | 0.97 (20.238)
  C5D1: number analyzed (Participants) | 56
  C5D1 | -0.89 (18.026)
  C6D1: number analyzed (Participants) | 52
  C6D1 | -1.92 (22.544)
  C7D1: number analyzed (Participants) | 34
  C7D1 | -5.39 (22.834)
  C8D1: number analyzed (Participants) | 27
  C8D1 | -4.63 (21.225)
  C9D1: number analyzed (Participants) | 18
  C9D1 | -1.85 (15.274)
  C10D1: number analyzed (Participants) | 13
  C10D1 | -7.69 (17.167)
  30 days safety Follow up: number analyzed (Participants) | 40
  30 days safety Follow up | -15.42 (25.775)

16. Secondary Outcome: Change From Baseline in EQ-5D-5L Over Time
Description: The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L VAS records the patient's self-rated health on a vertical visual analogue scale numbered from 0 ("The worst health you can imagine") to 100 ("The best health you can imagine"). Changes from baseline in EQ-5D-5L VAS over time are presented in this record.
Time Frame: From Cycle 1 Day 1 (C1D1) Visit to the 30-day Safety Follow-up Visit up to a maximum of 17.6 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Arm
Number analyzed (Participants) | 95
units on a scale
  C2D1: number analyzed (Participants) | 78
  C2D1 | 0.04 (19.707)
  C3D1: number analyzed (Participants) | 71
  C3D1 | 0.35 (21.668)
  C4D1: number analyzed (Participants) | 68
  C4D1 | 2.66 (19.400)
  C5D1: number analyzed (Participants) | 55
  C5D1 | 3.73 (17.052)
  C6D1: number analyzed (Participants) | 52
  C6D1 | 1.69 (18.421)
  C7D1: number analyzed (Participants) | 35
  C7D1 | 1.31 (18.903)
  C8D1: number analyzed (Participants) | 28
  C8D1 | 2.89 (15.882)
  C9D1: number analyzed (Participants) | 19
  C9D1 | -2.32 (21.945)
  C10D1: number analyzed (Participants) | 13
  C10D1 | -4.00 (12.503)
  30 days safety Follow up: number analyzed (Participants) | 40
  30 days safety Follow up | -9.35 (23.585)

17. Secondary Outcome: PGIC Scores Over Time
Description: The Patient Global Impression of Change (PGIC) is a measure of patients' perceptions of change in their symptoms over time. For this assessment, subjects answered the following question: "Since starting treatment, my colorectal cancer symptoms are: (1) very much improved, (2) much improved, (3) minimally improved, (4) no change, (5) minimally worse, (6) much worse or (7) very much worse."
Time Frame: From Cycle 1 Day 1 (C1D1) Visit to the 30-day Safety Follow-up Visit up to a maximum of 17.6 months
Population: PGIC scores are shown up to Cycle 10 Day 1 (C10D1) and for the 30-day safety follow-up period. Beyond C10D1, less than 10 subjects filled the questionnaire. Participants analyzed corresponds to the number of participant who completed the questionnaire the at the respective time point.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Arm
Number analyzed (Participants) | 95
Participants
  C2D1: number analyzed (Participants) | 91
  C2D1: Very much improved | 5
  C2D1: Much improved | 15
  C2D1: Minimally improved | 17
  C2D1: No change | 29
  C2D1: Minimally worse | 3
  C2D1: Much worse | 0
  C2D1: Very much worse | 0
  C2D1: Missing, not done | 22
  C3D1: number analyzed (Participants) | 81
  C3D1: Very much improved | 10
  C3D1: Much improved | 28
  C3D1: Minimally improved | 11
  C3D1: No change | 20
  C3D1: Minimally worse | 0
  C3D1: Much worse | 0
  C3D1: Very much worse | 0
  C3D1: Missing, not done | 12
  C4D1: number analyzed (Participants) | 77
  C4D1: Very much improved | 9
  C4D1: Much improved | 31
  C4D1: Minimally improved | 12
  C4D1: No change | 16
  C4D1: Minimally worse | 0
  C4D1: Much worse | 0
  C4D1: Very much worse | 0
  C4D1: Missing, not done | 9
  C5D1: number analyzed (Participants) | 65
  C5D1: Very much improved | 10
  C5D1: Much improved | 19
  C5D1: Minimally improved | 11
  C5D1: No change | 13
  C5D1: Minimally worse | 2
  C5D1: Much worse | 0
  C5D1: Very much worse | 0
  C5D1: Missing, not done | 10
  C6D1: number analyzed (Participants) | 57
  C6D1: Very much improved | 7
  C6D1: Much improved | 18
  C6D1: Minimally improved | 13
  C6D1: No change | 13
  C6D1: Minimally worse | 0
  C6D1: Much worse | 0
  C6D1: Very much worse | 0
  C6D1: Missing, not done | 6
  C7D1: number analyzed (Participants) | 43
  C7D1: Very much improved | 4
  C7D1: Much improved | 13
  C7D1: Minimally improved | 7
  C7D1: No change | 11
  C7D1: Minimally worse | 0
  C7D1: Much worse | 0
  C7D1: Very much worse | 0
  C7D1: Missing, not done | 8
  C8D1: number analyzed (Participants) | 33
  C8D1: Very much improved | 4
  C8D1: Much improved | 11
  C8D1: Minimally improved | 5
  C8D1: No change | 5
  C8D1: Minimally worse | 2
  C8D1: Much worse | 0
  C8D1: Very much worse | 0
  C8D1: Missing, not done | 6
  C9D1: number analyzed (Participants) | 20
  C9D1: Very much improved | 1
  C9D1: Much improved | 9
  C9D1: Minimally improved | 2
  C9D1: No change | 5
  C9D1: Minimally worse | 0
  C9D1: Much worse | 0
  C9D1: Very much worse | 0
  C9D1: Missing, not done | 3
  C10D1: number analyzed (Participants) | 14
  C10D1: Very much improved | 2
  C10D1: Much improved | 4
  C10D1: Minimally improved | 4
  C10D1: No change | 4
  C10D1: Minimally worse | 0
  C10D1: Much worse | 0
  C10D1: Very much worse | 0
  C10D1: Missing, not done | 0
  30 days safety Follow-up: number analyzed (Participants) | 72
  30 days safety Follow-up: Very much improved | 3
  30 days safety Follow-up: Much improved | 12
  30 days safety Follow-up: Minimally improved | 5
  30 days safety Follow-up: No change | 9
  30 days safety Follow-up: Minimally worse | 6
  30 days safety Follow-up: Much worse | 6
  30 days safety Follow-up: Very much worse | 0
  30 days safety Follow-up: Missing, not done | 31

ADVERSE EVENTS:
Time Frame: From patient enrolment date to 30 days after the last dose of study drug up to a maximum of 17.6 months
Description: Only treatment emergent Adverse Events are provided in summary tables. A treatment emergent adverse event (TEAE) is defined as any event that first occurred during the treatment period (i.e. from first treatment administration date up to last administration date + 30 days) or that worsened during that study period.
Arm/Group | 1 Arm
All-Cause Mortality (participants affected / at risk) | 27/95
Serious Adverse Events (participants affected / at risk) | 49/95
Other Adverse Events (participants affected / at risk) | 93/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Arm (N=95)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Detachment of retinal pigment epithelium (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 6 (6)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (5)
Subileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Diversion colitis (Injury, poisoning and procedural complications) | 1 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (8)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Arm (N=95)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 31 (43)
Abdominal pain upper (Gastrointestinal disorders) | 7 (11)
Amylase increased (Investigations) | 10 (17)
Anaemia (Blood and lymphatic system disorders) | 23 (60)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14)
Asthenia (General disorders) | 30 (67)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Blood creatine phosphokinase increased (Investigations) | 5 (7)
Blood creatinine increased (Investigations) | 9 (11)
Constipation (Gastrointestinal disorders) | 25 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 22 (36)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 38 (77)
Diarrhoea (Gastrointestinal disorders) | 64 (145)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (35)
Dysgeusia (Nervous system disorders) | 12 (13)
Dyspepsia (Gastrointestinal disorders) | 8 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (23)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Fatigue (General disorders) | 18 (38)
Flatulence (Gastrointestinal disorders) | 5 (5)
Headache (Nervous system disorders) | 10 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 6 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (9)
Insomnia (Psychiatric disorders) | 5 (6)
Lipase increased (Investigations) | 12 (24)
Mucosal inflammation (General disorders) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 42 (83)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (6)
Paronychia (Infections and infestations) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (16)
Pyrexia (General disorders) | 12 (19)
Rash (Skin and subcutaneous tissue disorders) | 38 (56)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (8)
Skin fissures (Skin and subcutaneous tissue disorders) | 11 (17)
Stomatitis (Gastrointestinal disorders) | 8 (16)
Vision blurred (Eye disorders) | 13 (17)
Vomiting (Gastrointestinal disorders) | 34 (59)
Weight decreased (Investigations) | 6 (8)

LIMITATIONS AND CAVEATS:
The absence of a comparator arm should be noted as a limitation. In addition, the short duration of the follow-up at the data cut-off date does not allow a robust estimate of OS results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03693170/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03693170/SAP_001.pdf